CLINICAL TRIAL: NCT06633159
Title: Register of Patients With Heart Failure Who Underwent Surgery to Correct Mitral Regurgitation by Percutaneous Catheter Implantation of MitraClip on the Mitral Valve.
Brief Title: MitraClip in Patients With Heart Failure
Acronym: MitraClip
Status: Recruiting | Type: Observational
Sponsor: The League of Clinical Research, Russia (Other)
Collaborators: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: СН-01-2023
Record Dates: First submitted 2024-09-23; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Mitral Regurgitation
Keywords: Clip implantation; Transcatheter plastic surgery; Mitral valve (MV); MitraClip; Mitral regurgitation (MR)
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- prospective: The prospective part of the study will include patients who have undergone hospitalization for the purpose of surgical intervention to correct mitral regurgitation by percutaneous transcatheter implantation of the MitraClip G4 clip on the mitral valve leaflets.
  Interventions: Device: MitraClip
- retrospective: The retrospective part of the study will include patients who underwent surgical intervention to correct mitral regurgitation by percutaneous transcatheter implantation of the MitraClip G4 clip on the mitral valve leaflets.
  Interventions: Device: MitraClip

INTERVENTIONS:
Device: MitraClip — surgical intervention to correct mitral regurgitation by percutaneous transcatheter implantation of the MitraClip G4 clip on the mitral valve leaflets

SUMMARY:
Multicenter observational study. The study does not involve any interventions in routine clinical practice, the choice of treatment method (including the type of medical device used and the method of surgical intervention) and the methods of examination and postoperative management of patients will not differ from the standard of care for patients requiring percutaneous transcatheter edge-to-edge mitral valve reconstruction by implantation of the MitraClip clip on the mitral valve leaflets, used in the daily medical practice of a medical institution. All medical devices under study (delivery device with the MitraClip clip on the mitral valve leaflets) are registered in the territory of the Russian Federation and are used in the conditions of routine medical practice. The study will include patients who have undergone surgical intervention to correct mitral regurgitation by percutaneous transcatheter implantation of the MitraClip G4 clip on the mitral valve leaflets. It is expected to include at least 196 patients (at least 98 prospective patients and at least 98 retrospective patients). The planned number of research centers is 11 outpatient clinics, presumably in 6 regions of the Russian Federation.

DETAILED DESCRIPTION:
Mitral regurgitation (MR) may result from either degenerative lesions of the mitral valve (MV) leaflets - degenerative MR (DMR) - or pathological dilation of the left ventricle (LV) - functional MR (FMR). In DMR, the MV apparatus itself is compromised by affected leaflets, chords, etc. In contrast, FMR is usually associated with cardiomyopathy (usually of ischemic etiology), with this type of MR being secondary to LV dysfunction. In both cases, there is a violation of leaflet co-optation and reverse blood flow from the LV into the left atrium. According to existing guidelines, surgical reconstruction (plastic surgery) is the preferred treatment option for DMR. Indications for invasive treatment of FMR are not so clear-cut due to the high rate of postoperative MR recurrence and the lack of reliable evidence of a positive effect of FMR correction on long-term survival. The greatest complexity is presented by the group of patients with severe MR and high or unacceptable surgical risk of open surgery.

For the treatment of severe MR in such patients, the method of transcatheter MV repair was proposed, which is an endovascular analogue of the suture "edge-to-edge" repair according to Alfieri. MitraClip system is approved in the European Union, the USA, the Middle East and the CIS (Kazakhstan, Belarus) for the treatment of high surgical risk patients with DMR and FMR with symptomatic heart failure of II-IV functional class according to the classification of the New York Heart Association (NYHA), persisting despite optimal drug therapy.

The aim of this study is to evaluate the safety and effectiveness of the procedure of percutaneous transcatheter implantation of the MitraClip G4 clip on the mitral valve leaflets in a population of patients from the Russian Federation for the treatment of mitral regurgitation. Information on the health status of patients who have undergone the procedure of percutaneous transcatheter edge-to-edge mitral valve reconstruction by implanting the MitraClip clip on the mitral valve leaflets will be of high scientific and practical interest.

ELIGIBILITY:
Cohort 1 (prospective patients)

Inclusion Criteria:

1. Patients who are indicated for cardiac surgery to correct mitral regurgitation using transcatheter edge-to-edge reconstruction of the mitral valve by implanting the MitraClip G4 on the cusps of the mitral valve.
2. Age 18 years and older.
3. Understanding and voluntarily signing the informed consent form for the processing of personal data.

Exclusion Criteria:

1. The expected life expectancy of the patient is less than 12 months (contraindication to surgical intervention).
2. The presence of concomitant diseases that limit the patient's ability to carry out visits according to the study protocol.
3. Conditions that limit the patient's ability to comply with the study requirements (dementia, psychoneurological diseases, drug addiction, alcoholism, etc.).
4. Simultaneous participation in other clinical trials or previous participation in this trial.

Cohort 2 (retrospective patients)

Inclusion Criteria:

1.Patients who underwent cardiac surgery to correct mitral regurgitation using transcatheter edge-to-edge mitral valve reconstruction with MitraClip G4 clip implantation on the mitral valve leaflets.

Exclusion Criteria:

1. Patients for whom the physician-researcher cannot access primary medical documentation (medical records, outpatient cards) to collect complete and reliable information about the patient in the volume required by the study protocol.
2. The surgery must have been performed no earlier than January 1, 2022.
3. Age 18 years and older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older with heart failure and implanted MitraClip G4 mitral valve clips.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | Month 12
  To evaluate cardiovascular mortality within 12 months in patients with heart failure after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.

SECONDARY OUTCOMES:
All-cause mortality | Month 12
  To assess all-cause mortality within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Hospitalization for heart failure | Month 12
  To assess the incidence of hospitalization for heart failure within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Hospitalization for any cause | Month 12
  To assess the incidence of hospitalization for any cause within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Emergency surgical interventions | Month 12
  To assess the frequency of unplanned (emergency) surgical interventions on the mitral valve within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Functional class of heart failure | Month 1 - Month 3 - Month 12
  To assess the change in the functional class of heart failure within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
N-terminal pre-brain natriuretic peptide | Month 1 - Month 12
  To assess the change in the level of N-terminal pre-brain natriuretic peptide over 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Echocardiographic examination: severity of mitral regurgitation: I-IV; | Month 1 - Month 12
  To evaluate the change in echocardiographic examination parameters within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Echocardiographic examination:presence of severe mitral valve stenosis ; | Month 1 - Month 12
  To evaluate the change in echocardiographic examination parameters: presence of severe mitral valve stenosis within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Surgical complications | Month 12
  To assess the incidence of surgical complications within 12 months after correction of mitral regurgitation by percutaneous transcatheter implantation of the MitraClip on the mitral valve leaflets.
Safety of surgical intervention | Month 12
  Surgical complications after correction of mitral regurgitation: yes/no. If yes: date of development of the complication, description of the complication (ICD-10 term), outcome of the complication at the 12-month follow-up period (death, resolved without consequences, resolved with consequences, ongoing).
Safety of surgical intervention:AE | Month 12
  Adverse events: yes/no If yes: date of development of the AE, description of the AE (ICD-10 term), outcome of the AE by the 12-month follow-up period (death, resolved without consequences, resolved with consequences, ongoing).
Safety of surgical intervention: сardiac surgery | Month 12
  Cardiac surgery during the 12-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Sergey A Boytsov, Prof., Study Chair — Research Institute of Cardiology
Locations (1):
- League of Clinical Research (LeagueCRR), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No